CLINICAL TRIAL: NCT00093353
Title: A Phase I Study Of Oral Irinotecan, Temozolomide, Cefixime In Children With Recurrent/Resistant High-Risk Neuroblastoma
Brief Title: N2003-01: Irinotecan, Temozolomide, and Cefixime in Treating Young Patients With Recurrent or Resistant Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Lars Wagner, M.D., Cincinnati Children's Hospital Medical Center
Purpose: Treatment
Other Study IDs: CDR0000373759; P01CA081403 (NIH); N2003-01 (Other: NANT Consortium)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2009-05

CONDITIONS: Diarrhea; Drug/Agent Toxicity by Tissue/Organ; Neuroblastoma
Keywords: diarrhea; drug/agent toxicity by tissue/organ; disseminated neuroblastoma; recurrent neuroblastoma
MeSH Terms: conditions — Diarrhea; Drug-Related Side Effects and Adverse Reactions; Neuroblastoma | interventions — Cefixime; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cefixime
Drug: irinotecan hydrochloride
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Temozolomide may help irinotecan kill more tumor cells by making them more sensitive to the drug. Cefixime may be effective in preventing diarrhea that is caused by treatment with irinotecan.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan when given together with temozolomide and cefixime in treating young patients with recurrent or resistant neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of oral irinotecan when administered with fixed-dose temozolomide and cefixime in pediatric patients with recurrent or resistant high-risk neuroblastoma.
* Determine the toxic effects of this regimen in these patients.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.
* Correlate UGT1A1 genotype with the occurrence of dose-limiting diarrhea in patients treated with this regimen.
* Correlate BCRP genotype with pharmacokinetic phenotype in patients treated with this regimen.
* Correlate p53 status in tumor cells with response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of irinotecan.

Patients receive oral cefixime once daily beginning 5 days before the start of fixed-dose temozolomide and irinotecan and continuing for the duration of the study. Patients also receive oral temozolomide once daily on days 1-5 and oral irinotecan once daily on days 1-5 and 8-12. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A maximum of 12 patients are treated at the MTD.

Patients are followed for toxicity, response, and survival.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 1.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma AND/OR demonstration of tumor cells in the bone marrow with increased urinary catecholamines

  * High-risk disease meeting 1 of the following criteria:

    * Recurrent or progressive disease
    * Resistant or refractory disease (i.e., never achieved a complete response to therapy AND never had new sites of disease or progression of initial sites)
* Measurable disease meeting at least 1 of the following criteria:

  * Unidimensionally measurable tumor ≥ 20 mm by MRI, CT scan, or x-ray OR ≥ 10 mm by spiral CT scan*
  * At least 1 site with positive uptake by metaiodobenzylguanidine (MIBG) scan*
  * Bone marrow with tumor cells seen on routine morphology (not by NSE staining only) of bilateral aspirate AND/OR biopsy on 1 bone marrow sample NOTE: *Patients who never experienced disease recurrence or progression must demonstrate viable neuroblastoma in a biopsy of either bone marrow or bone and/or soft tissue site (biopsy must be performed ≥ 4 weeks after completion of prior radiotherapy if lesion was irradiated)

PATIENT CHARACTERISTICS:

Age

* 1 to 30 at diagnosis

Performance status

* ECOG 0-2

Life expectancy

* At least 2 months

Hematopoietic

* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3 (without transfusion)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)

Hepatic

* SGPT and SGOT < 5 times normal
* Bilirubin ≤ 1.5 times normal

Renal

* Creatinine ≤ 1.5 times normal for age

  * No greater than 0.8 mg/dL (≤ 5 years of age)
  * No greater than 1.0 mg/dL (6 to 10 years of age)
  * No greater than 1.2 mg/dL (11 to 15 years of age)
  * No greater than 1.5 mg/dL (> 15 years of age)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to cephalosporins
* No active diarrhea
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* Recovered from prior immunotherapy
* More than 3 weeks since prior biologic therapy and recovered
* More than 2 days since prior hematopoietic growth factors
* No concurrent epoetin alfa
* No concurrent prophylactic hematopoietic growth factors during the first treatment course
* No concurrent immunomodulating agents except steroids to control intracranial pressure

Chemotherapy

* Prior myeloablative therapy and autologous stem cell transplantation allowed

  * No prior allogeneic stem cell transplantation
* More than 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* Prior temozolomide, irinotecan, or topotecan allowed

  * No prior temozolomide and irinotecan as combination therapy
* No other concurrent chemotherapy

Endocrine therapy

* See Biologic therapy

Radiotherapy

* At least 6 weeks since prior large field radiotherapy (e.g., total body irradiation, craniospinal therapy, whole abdomen, total lung, or > 50% bone marrow space) and recovered
* At least 4 weeks since prior radiotherapy to biopsied lesions (for study entry) and recovered
* At least 6 weeks since prior MIBG therapy
* Concurrent radiotherapy to painful lesions allowed provided the lesions are not used to assess treatment response

Surgery

* Not specified

Other

* No concurrent enzyme-inducing anticonvulsants (e.g., phenobarbital, phenytoin, or carbamazepine)
* No other concurrent anticancer agents

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars M. Wagner, MD, Study Chair — Children's Hospital Medical Center, Cincinnati; Katherine K. Matthay, MD, Principal Investigator — University of California, San Francisco
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Wagner LM, Villablanca JG, Stewart CF, Crews KR, Groshen S, Reynolds CP, Park JR, Maris JM, Hawkins RA, Daldrup-Link HE, Jackson HA, Matthay KK. Phase I trial of oral irinotecan and temozolomide for children with relapsed high-risk neuroblastoma: a new approach to neuroblastoma therapy consortium study. J Clin Oncol. 2009 Mar 10;27(8):1290-6. doi: 10.1200/JCO.2008.18.5918. Epub 2009 Jan 26. PMID 19171709